CLINICAL TRIAL: NCT00087152
Title: Phase II Trial Of Imatinib Mesylate (Gleevec®) (NSC-716051) In Combination With Capecitabine (Xeloda®) (NSC-712807) In Metastatic Breast Cancer
Brief Title: S0338, Imatinib Mesylate and Capecitabine in Treating Women With Progressive Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03033; U10CA032102 (NIH); S0338 (Other: SWOG); CDR0000372950 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate & Capecitabine (Experimental)
  Interventions: Drug: Capecitabine; Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Capecitabine — 1,000 mg/m^2 by mouth twice daily Days 1-14 of each 21 day cycle
  Other Names: Xeloda
Drug: Imatinib mesylate — 400 mg by mouth daily
  Other Names: Gleevec

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining imatinib mesylate with capecitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving imatinib mesylate together with capecitabine works in treating women with progressive stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the confirmed complete and partial response rate in women with progressive stage IV adenocarcinoma of the breast treated with imatinib mesylate and capecitabine.
* Determine the 6-month progression-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Correlate, preliminarily, c-kit and platelet-derived growth factor receptor expression with estrogen and progesterone receptor status, response, survival, and time to disease progression in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate* once daily on days 1-21 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *If the patient tolerates the starting dose of imatinib mesylate in course 1, the dose will be increased in subsequent courses.

Patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 25-70 patients (25-45 patients with measurable disease and 25 with non-measurable disease) will be accrued for this study within 2 years.

ELIGIBILITY:
* Histologically or cytologically confirmed adenocarcinoma of the breast
* Stage IV measurable disease
* Disease progression after at least 1, but no more than 2, prior chemotherapy regimens for metastatic disease
* Patients with hormone-sensitive tumors must have received prior hormonal therapy
* Patients with human epidermal growth factor receptor 2 (HER2)/neu-overexpressing tumors (3+ by immunohistochemistry or amplified by fluorescent in situ hybridization) should have received trastuzumab (Herceptin®) in the adjuvant or metastatic setting (unless contraindicated)
* No clinical evidence of or known brain or central nervous system (CNS) disease
* Hormone Receptor status known
* Female age 18 and over
* Performance status Zubrod 0-2
* Absolute neutrophil count > 1,500/mm^3
* Leukocyte count > 3,000/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin normal
* aspartate aminotransferase (AST) / alanine aminotransferase (ALT) < 2.5 times upper limit of normal
* Creatinine normal OR Creatinine clearance > 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation
* No history of severe hypersensitivity reaction to compounds of similar chemical or biological composition to imatinib mesylate, capecitabine, or fluorouracil
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No prior biologic therapy (e.g., vaccines)
* No concurrent filgrastim (G-CSF) for chemotherapy-induced neutropenia
* No prior capecitabine or fluorouracil for metastatic breast cancer
* Prior hormonal therapy allowed
* More than 4 weeks since prior radiotherapy - Previously irradiated area(s) must not be the only site of disease
* More than 4 weeks since prior major surgery
* More than 4 weeks since prior therapy for breast cancer
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for metastatic breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen K. Chew, MD, Study Chair — University of California, Davis; Kathy S. Albain, MD, Study Chair — Loyola University

REFERENCES:
- [Result] Chew HK, Barlow WE, Albain K, Lew D, Gown A, Hayes DF, Gralow J, Hortobagyi GN, Livingston R. A phase II study of imatinib mesylate and capecitabine in metastatic breast cancer: Southwest Oncology Group Study 0338. Clin Breast Cancer. 2008 Dec;8(6):511-5. doi: 10.3816/CBC.2008.n.062. PMID 19073506
- [Result] Chew HK, Barlow W, Albain K, et al.: SWOG 0338: a phase II trial of imatinib mesylate in combination with capecitabine in metastatic breast cancer. [Abstract] J Clin Oncol 24 (Suppl 18): A-10529, 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated June 15, 2004. It was open to SWOG institutions who obtained Institutional Review Board (IRB) approval for this study. 27 patients were enrolled at 16 institutions. The study was temporarily closed to accrual April 19, 2005 to allow assessment of response in the first stage. It was closed permanently on December 15, 2005.
Groups:
- Imatinib Mesylate & Capecitabine: Imatinib Mesylate 400 mg by mouth daily for 21 day cycle. Capecitabine 1,000 mg/m^2 by mouth twice daily Days 1-14 of each 21 day cycle.
Period: Overall Study
Arm/Group | Imatinib Mesylate & Capecitabine
Started | 27
Completed | 21
Not Completed | 6
Not completed — Ineligible | 6

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate & Capecitabine
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Complete and Partial)
Description: Number of participants with confirmed complete or partial response. Confirmed response (complete and partial) per Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (V1.0). Complete Response (CR) is complete disappearance of all measurable and non-measurable disease; no new lesions; no disease related symptoms; and normalization of markers and other abnormal lab values. Partial response (PR) applies only to patients with at least one measurable lesion. PR is greater than or equal to 30% decrease under baseline of the sum of longest diameter of all target measurable lesions; no unequivocal progression of non-measurable disease and no new lesions. Confirmed response is two or more objective statuses a minimum of four weeks apart documented before progression or symptomatic deterioration.
Time Frame: 12 weeks
Population: Eligible participants who received treatment.
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate & Capecitabine
Number analyzed (Participants) | 19
participants | 2

2. Secondary Outcome: Progression-free Survival at 6 Months
Description: Percentage of participants progression-free at 6 months. Progression-free survival (PFS) measured from date of registration to first observation of progressive disease (per RECIST criteria (V1.0)), death due to any cause, or symptomatic deterioration. Kaplan-Meier was used to estimate progression-free survival (PFS) at six months.
Time Frame: Six months
Population: Eligible participants who received treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate & Capecitabine
Number analyzed (Participants) | 19
percentage of participants | 16 [0 to 32]

3. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5= Fatal. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Every 3 weeks while on treatment for up to 3 years.
Population: Eligible participants who received any treatment.
Measure: Number; unit: Participants
Groups:
- Imatinib Mesylate and Capecitabine: Imatinib Mesylate 400 mg by mouth daily for 21 day cycle. Capecitabine 1,000 mg/m^2 by mouth twice daily Days 1-14 of each 21 day cycle.
Arm/Group | Imatinib Mesylate and Capecitabine
Number analyzed (Participants) | 20
Participants
  Diarrhea | 2
  Fatigue (asthenia, lethargy, malaise) | 2
  Leukocytes (total WBC) | 1
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1
  Neuropathy: motor | 1
  Neuropathy: sensory | 1
  Neutrophils/granulocytes (ANC/AGC) | 1
  Pain - Abdomen NOS | 1
  Pain - Muscle | 1
  Rash/desquamation | 1
  Rash: hand-foot skin reaction | 2

ADVERSE EVENTS:
Time Frame: Every 3 weeks while on treatment for up to 3 years.
Arm/Group | Imatinib Mesylate and Capecitabine
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate and Capecitabine (N=20)
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate and Capecitabine (N=20)
Hemoglobin (Blood and lymphatic system disorders) | 14
Ocular/Visual-Other (Specify) (Eye disorders) | 1
Optic disc edema (Eye disorders) | 1
Watery eye (epiphora, tearing) (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 7
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 14
Pain - Abdomen NOS (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Death not associated with CTCAE term - Death NOS (General disorders) | 1
Edema: head and neck (General disorders) | 2
Edema: limb (General disorders) | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 15
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 2
AST, SGOT (Investigations) | 2
Alkaline phosphatase (Investigations) | 3
Bilirubin (hyperbilirubinemia) (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 9
Platelets (Investigations) | 5
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 5
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Dizziness (Nervous system disorders) | 2
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 4
Ocular/Visual-Other (Specify) (Nervous system disorders) | 1
Pain - Head/headache (Nervous system disorders) | 2
Taste alteration (dysgeusia) (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mood alteration - anxiety (Psychiatric disorders) | 1
Mood alteration - depression (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6
Flushing (Vascular disorders) | 1
Hot flashes/flushes (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Two-stage design, but did not have enough confirmed responses after the first stage to launch the second stage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less